CLINICAL TRIAL: NCT02522767
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study Investigating the Efficacy and Safety of Mesalamine 4 g Extended Release Granules (Sachet) for the Induction of Clinical and Endoscopic Remission in Active, Mild to Moderate Ulcerative Colitis
Brief Title: Mesalamine 4 g Sachet for the Induction of Remission in Active, Mild to Moderate Ulcerative Colitis (UC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 000174; 2015-002557-35 (EudraCT Number)
Record Dates: First submitted 2015-08-12; First posted 2015-08-13 (Estimated); Results first posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesalamine (Experimental): 4 g extended release granules (sachet)
  Interventions: Drug: Mesalamine
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mesalamine
  Other Names: Mesalazine; Pentasa
  Arms: Mesalamine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this trial is to investigate the efficacy of mesalamine for the induction of clinical and endoscopic remission in subjects with active, mild to moderate UC. Subject will receive 4 g extended release granules (sachet) once daily.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 to 75 years
* Mild to moderate UC

Exclusion Criteria:

* Disease limited to proctitis <15 cm
* Short bowel syndrome
* Prior colon resection surgery
* History of severe/fulminant UC
* Evidence of other forms of inflammatory bowel disease
* Infectious disease (including human immunodeficiency virus [HIV], hepatitis B virus [HBV], or hepatitis C virus [HCV])
* Intolerant or allergic to aspirin or salicylate derivatives
* Use of rectal formulations (5-aminosalicylic acid [5-ASA], steroids) within ≤7 days
* Women who are pregnant or nursing
* History or known malignancy
* History of bleeding disorders, active gastric or active duodenal ulcers, autoimmune diseases, or mental/emotional disorders, that would interfere with their participation in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (93):
- United States (18):
  - Preferred Research Partners, Little Rock, Arkansas
  - United Research Institute, Murrieta, California
  - Research Associates of South Florida, LLC, Miami, Florida
  - IMIC, Palmetto Bay, Florida
  - Medical Research Center of Florida, Pembroke Pines, Florida
  - Lenus Research and Medical Group, Sweetwater, Florida
  - Clinical Trials of SWLA, LLC, Lake Charles, Louisiana
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Wilmington Gastroenterology Associates, Wilmington, North Carolina
  - Associates in Gastroenterology, PLC, Hermitage, Tennessee
  - Quality Medical Research, PLLC, Nashville, Tennessee
  - BI Research Center, Houston, Texas
  - Biopharma Informatic Inc., Houston, Texas
  - Digestive Health Center, Pasadena, Texas
  - DM Clinical Research, Tomball, Texas
  - Advanced Research Institute, Ogden, Utah
  - New River Valley Research Institute, Christiansburg, Virginia
  - Digestive & Liver Disease Specialists, Norfolk, Virginia
- Bulgaria (8):
  - Multiprofile Hospital For Active Treatment Avis Medica, Pleven
  - Medical Center Excelsior OOD, Sevlievo
  - Medical Center-1-Sevlievo EOOD, Sevlievo
  - City Clinic University Multiprofile Hospital for Active Treatment EOOD, Sofia
  - Medical Center Asklepion - Humane Medicine Research EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment Sv Ivan Rilski EAD, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna - ISUL EAD, Sofia
  - Diagnostic Consultative Centre Mladost M OOD, Varna
- Canada (2):
  - Topstone Research Institute, Ottawa, Ontario
  - Toronto Digestive Disease Associates, Vaughan
- Hungary (7):
  - Magyar Honvédség Egészségügyi Központ, Budapest
  - Pannónia Magánorvosi Centrum Kft, Budapest
  - Semmelweis Egyetem Institute, Budapest
  - Vasútegészségügyi Nonprofit Kiemelten Közhasznú Kft. Debreceni Egészségügyi Központja, Debrecen
  - ENDOMEDIX Kft., Miskolc
  - Karolina Korhaz Rendelointezet, Mosonmagyaróvár
  - Clinfan Kft., Szekszárd
- Latvia (5):
  - Polana-D, LTD, Daugavpils
  - Digestive Diseases Centre Gastro, Riga
  - Latvian Maritime Medicine Centre, Riga
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga East Clinical University Hospital, Riga
- Mexico (3):
  - ICARO Investigaciones en Medicina, S.A de C.V, Chihuahua City
  - Maria Auxiliadora Hospital, Guadalajara
  - Investigación Biomédica para el Desarrollo de Fármacos, S.A. de C.V., Zapopan
- Poland (12):
  - Osrodek Medycyny Rodzinnej Sp. z o.o., Sobótka, Lower Silesian Voivodeship
  - Lexmedica, Wroclaw, Lower Silesian Voivodeship
  - Zespół Przychodni Specjalistycznych PRIMA Sp. z o.o., Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej Intermed, Częstochowa
  - Economicus - NZOZ ALL-MEDICUS, Katowice
  - Investigational site, Ksawerów
  - Niepubliczny Zaklad Opieki Zdrowotnej CENTRUM MEDYCZNE Szpital Swietej Rodziny, Lodz
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
  - Investigational site, Sopot
  - Centrum Zdrowia Matki, Dziecka i Mlodziezy, Warsaw
- Russia (13):
  - Regional Clinical Hospital, Krasnoyarsk
  - City Clinical Hospital #51, Moscow
  - Nizhegorodskaya Regional Clinical Hospital n.a. Semashko, Nizhny Novgorod
  - Novosibirsk State Medical University, Novosibirsk
  - Research Institute of Physiology of Sibirian Branch the RAMS, Novosibirsk
  - Omsk State Medical Academy, Omsk
  - Rostov State Medical University, Rostov-on-Don
  - State Budget Institution of Ryazan region" Regional Clinical Hospital", Ryazan
  - City Hospital #31, Saint Petersburg
  - City Polyclinic #38, Saint Petersburg
  - Russian Medical Military Academy n.a. S.M. Kirov, Saint Petersburg
  - Railway Clinical Hospital at Station Samara OAO Rzhd, Samara
  - Stavropol State Medical Academy, Stavropol
- Serbia (2):
  - Clinical Hospital Centar Zvezdara, Belgrade
  - Health Center Valjevo, Valjevo
- Switzerland (3):
  - Inselspital Bern, Bern
  - Investigational site, Bern
  - Universitätsspital Zürich, Zurich
- Ukraine (20):
  - Kyiv Municipal Clinical Hospital #18, Kyiv, Kyïv
  - Medical Center LLC Ukrainian German Antiulcer Gastroenterology Center BIK Kyiv, Kyiv, Kyïv
  - Regional Municipal Institution Chernivtsi Regional Clinical Hospital, Chernivtsi
  - Municipal Institution Dnipropetrovsk Regional Clinical Hospital n.a. I.I. Mechnykov, Dnipropetrovsk
  - Municipal Healthcare Institution Kharkiv City Clinical Hospital #2, Kharkiv
  - SI National Institute of Therapy n.a. L.T. Mala of National Academy of Medical Sciences of Ukraine, Kharkiv
  - Municipal Intitution "Kherson City Clinical Hospital n.a. A. and O. Tropinykh", Kherson
  - Private Enterprise Private Manufactire Company "Acinus"., Kirovohrad
  - Kremenchuk city Hospital # n.a O.T.Bohaievskyi, Kremenchuk
  - Kyiv City Clinical Hospital #8, Kyiv
  - Kyiv Municipal Clinical Hospital #18, Kyiv
  - Medical Center Universal Clinic Oberih of LLC Kapytal, Kyiv
  - Municipal City Clinical emergency Hospital, Lviv
  - Municipal Institution Odesa Regional Clinical Hospital, Odesa
  - Medical Clinical Research Center of Medical Center LLC Health Clinic, Vinnytsia
  - Small Business Private Enterprise Medical Center "Pulse", Vinnytsia
  - Vinnytsia Regional Clinical Hospital Hospital n.a. M.I. Pyrohov, Vinnytsia
  - Municipal Institution 6th City Clinical Hospital of Zaporizhzhia City Council, Zaporizhzhia
  - Municipal Institution Zaporizhzhia Regional Clinical Hospital of Zaporizhzhia Regional Council, Zaporizhzhia
  - Medical Centre of PE First Private Clinic, Zhytomyr

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 71 sites in 10 countries (Bulgaria, Canada, Hungary, Latvia, Mexico, Russia, Serbia, Switzerland, Ukraine, and United States) recruited subjects to this trial between October 2015 to November 2017, the last subject completed last visit in April 2018.
Pre-assignment Details: A total of 411 subjects were screened, of which 228 subjects were randomized in a 1:1 ratio to either mesalamine or placebo group (114 subjects each), for 8 weeks double-blind treatment.
  Subjects who completed 8 weeks but failed to meet the defined criteria for remission received open-label treatment with mesalamine for additional 8 weeks.
Groups:
- Mesalamine: Mesalamine 4 gram (g) extended release granules (sachet), administered orally once daily (QD)
- Placebo: Placebo 4 g to match mesalamine extended release granules, administered orally QD
Period: Double-blind
Arm/Group | Mesalamine | Placebo
Started | 114 | 114
Completed | 103 | 90
Not Completed | 11 | 24
Not completed — Withdrawal by Subject | 8 | 11
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 1 | 10
Not completed — Protocol Violation | 0 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Protocol Deviation | 1 | 0
Period: Open-label
Arm/Group | Mesalamine | Placebo
Started | 88 (Subjects provided their consent to receive additional 8 weeks open-label treatment with mesalamine.) | 82 (Subjects provided their consent to receive additional 8 weeks open-label treatment with mesalamine.)
Completed | 83 | 75
Not Completed | 5 | 7
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intention-to-treat (ITT) analysis set comprised all randomized subjects.
Groups:
- Mesalamine: Mesalamine 4 g extended release granules (sachet), administered orally QD
- Total: Total of all reporting groups
Arm/Group | Mesalamine | Placebo | Total
Number analyzed (Participants) | 114 | 114 | 228
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 107 | 105 | 212
  >=65 years | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (13.09) | 43.9 (13.68) | 42.5 (13.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 64 | 121
  Male | 57 | 50 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 18
  Not Hispanic or Latino | 105 | 105 | 210
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 5 | 8
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 105 | 103 | 208
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.68 (4.546) | 24.63 (4.578) | 24.66 (4.552)
Stool Frequency Score [Mean (Standard Deviation); unit: scores on a scale] — Stool Frequency Score is graded 0-3, where 0 is best.
  scores on a scale | 1.6 (0.81) | 1.8 (0.78) | 1.7 (0.80)
Rectal Bleeding Score [Mean (Standard Deviation); unit: scores on a scale] — Rectal Bleeding Score is graded 0-3, where 0 is best.
  scores on a scale | 1.2 (0.54) | 1.2 (0.58) | 1.2 (0.55)
Endoscopic Response Score [Mean (Standard Deviation); unit: scores on a scale] — Endoscopic Response Score is graded 0-3, where 0 is best.
  scores on a scale | 2.7 (0.47) | 2.6 (0.48) | 2.7 (0.47)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Remission
Description: The proportion of subjects with remission was defined by the Clinical and Endoscopic Response Score: 0 for rectal bleeding; 0 or 1 with at least 1 point decrease from baseline for stool frequency; 0 or 1 for endoscopic score.
  The Clinical and Endoscopic Response Score ranged between 0-9, higher scores indicating greater disease severity. This score had two components: Clinical Response which assessed subject's symptoms and ranged between 0-6, and Endoscopic Response which assessed objective evidence of inflammation and ranged between 0-3.
  Further, the Clinical Response component included two subscales: stool frequency and rectal bleeding (each ranged between 0-3 each) obtained from subjects' daily records. The Endoscopic Response component had one subscale: flexible sigmoidoscopy/colonoscopy (ranging between 0-3).
Time Frame: At Week 8
Population: The ITT analysis set comprised all randomized subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 114 | 114
Participants | 19 | 13
Statistical Analysis 1: Comparison: Mesalamine vs Placebo; Proportions were compared between treatment groups, at a two-sided 0.05 significance level; Test type: Superiority; p > 0.05, Chi-squared — The p-value was based on chi-square test without a continuity correction; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.73 to 3.32]

2. Secondary Outcome: Proportion of Subjects With Remission in the Primary Endpoint and the Physician's Global Assessment (PGA) Score of ≤1 (Modified Mayo Score)
Description: The Modified Mayo score was calculated as the sum of the Clinical and Endoscopic Response Score (Range: 0-9, and the standard PGA score (range: 0-3; normal [score=0], mild disease [score=1], moderate disease [score=2], severe disease [score=3]).
  The statistical test was to be conducted only if the primary analysis was significant.
Time Frame: At Week 8
Population: The ITT analysis set comprised all randomized subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 114 | 114
Participants | 19 | 11

3. Secondary Outcome: Time to Cessation of Rectal Bleeding
Description: Defined as time in days from randomization to the first day of 3 consecutive days with a rectal bleeding score of 0, based on subject's daily diary.
  The statistical test was to be conducted only if the primary analysis was significant.
Time Frame: Up to Week 8
Population: The ITT analysis set comprised all randomized subjects.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 114 | 114
days | 18.0 [13.0 to 30.0] | 43.0 [23.0 to NA] — Not estimable: Not estimable due to insufficient number of participants with cessation.

4. Secondary Outcome: The Proportion of Subjects With Endoscopic Improvement
Description: Defined as an Endoscopic Response Score of 0 or 1, with at least a 1 point reduction from baseline in the endoscopic score at Week 8.
Time Frame: At Week 8
Population: The ITT analysis set comprised randomized subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 114 | 114
Participants | 34 | 22
Statistical Analysis 1: Comparison: Mesalamine vs Placebo; Proportions were compared between treatment groups at a two-sided 0.05 significance level; Test type: Superiority; p > 0.05, Chi-squared — The p-value was based on chi-square test without a continuity correction; Odds Ratio (OR) = 1.78, 95% CI 2-sided [0.96 to 3.29]

5. Secondary Outcome: The Proportion of Subjects in Clinical Remission at Weeks 2, 4, and 8
Description: Defined as a score of 0 for rectal bleeding and 0 or 1 with at least 1 point decrease from baseline for stool frequency in the Clinical Response Score subset.
Time Frame: At Week 2, 4, and 8
Population: The ITT analysis comprised all randomized subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 114 | 114
Participants
  Week 2 | 19 | 17
  Week 4 | 29 | 26
  Week 8 | 40 | 28
Statistical Analysis 1: Comparison: Mesalamine vs Placebo; Proportions were compared between treatment groups over 8 weeks, at a two-sided 0.05 significance level; Test type: Superiority; p > 0.05, Generalized estimating equation approach; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.78 to 2.15]

6. Secondary Outcome: Time to Normal Stool Pattern
Description: Defined as time in days from randomization to the first day of 3 consecutive days with a stool frequency score of 0, based on subject daily diary.
Time Frame: Up to Week 8
Population: The ITT analysis set comprised randomized subjects.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 114 | 114
days | 55.0 [35.0 to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Mesalamine vs Placebo; Times to normal stool pattern were compared between treatment groups, at a two-sided 0.05 significance level; Test type: Superiority; p > 0.05, Log Rank — The p-value was based on log-rank test; Hazard Ratio (HR) = 1.36, 95% CI 2-sided [0.91 to 2.02] — Hazard ratio and its 95% CI were obtained from Cox proportional hazards model with treatment group as a factor

7. Secondary Outcome: The Change From Baseline in Rectal Bleeding Score at Weeks 2, 4, and 8
Description: Defined as change from baseline in rectal bleeding score at Week 2, 4, and 8 based on subject daily diary. Rectal Bleeding Score is graded 0-3, where 0 is best.
Time Frame: From baseline to Week 2, 4, and 8
Population: The ITT analysis set comprised randomized subjects.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 114 | 114
scores on a scale
  Week 2 | -0.39 (0.68) | -0.23 (0.84)
  Week 4 | -0.56 (0.72) | -0.34 (0.92)
  Week 8 | -0.64 (0.80) | -0.35 (0.84)
Statistical Analysis 1: Comparison: Mesalamine vs Placebo; Change from baseline scores were compared between treatment groups over 8 weeks, at a two-sided 0.05 significance level; Test type: Superiority; p < 0.05, Repeated-measures ANCOVA; Treatment difference = -0.24, 95% CI 2-sided [-0.41 to -0.08] — A repeated-measures ANCOVA model with an unstructured correlation matrix was used to calculate estimate

8. Secondary Outcome: The Change From Baseline in Serum C-reactive Protein (CRP) Levels at Weeks 2, 4, and 8
Description: The adjusted mean changes in serum CRP levels from baseline and their difference between treatment groups are presented for each time point.
Time Frame: From baseline to Week 2, 4, and 8
Population: The ITT analysis set comprise all randomized subjects.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 114 | 114
mg/L
  Week 2 | 0.60 (13.52) | 0.25 (19.67)
  Week 4 | -0.86 (16.52) | -1.05 (16.27)
  Week 8 | -2.01 (13.09) | -0.73 (22.51)
Statistical Analysis 1: Comparison: Mesalamine vs Placebo; Change from baseline scores were compared between treatment groups over 8 weeks, at a two-sided 0.05 significance level; Test type: Superiority; p > 0.05, Repeated-measures ANCOVA; Treatment difference = -2.39, 95% CI 2-sided [-5.46 to 0.67] — A repeated-measures ANCOVA model with an unstructured correlation matrix was used to calculate estimate

9. Secondary Outcome: The Change From Baseline in Fecal Calprotectin Levels at Week 8
Description: The adjusted mean change from baseline in fecal calprotectin levels at Week 8 are presented.
Time Frame: From baseline to Week 8
Population: The ITT analysis set comprised all randomized subjects.
Measure: Mean (Standard Deviation); unit: ug/g
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 114 | 114
ug/g | -144.93 (854.41) | -119.56 (1083.69)
Statistical Analysis 1: Comparison: Mesalamine vs Placebo; Changes from baseline were compared between treatment groups, at a two-sided 0.05 significance level; Test type: Superiority; p < 0.05, ANCOVA; Treatment difference = -289.69, 95% CI 2-sided [-514.96 to -64.42] — An ANCOVA model was used to calculate estimates

10. Secondary Outcome: The Change From Baseline in Health Related Quality of Life (QoL) Scores
Description: The change from baseline to Week 2, 4, and 8 in Inflammatory Bowel Disease Questionnaire (IBDQ) scores.
  The adjusted changes from baseline and their differences between treatment groups are presented.
  The IBDQ is an instrument used to assess quality of life in adult patients with UC.
  Subjects were asked to recall symptoms and QoL from last two weeks and to rate each item on a 7- point Likert score (higher scores equate to higher QoL).
Time Frame: From baseline to Week 2, 4, and 8
Population: The ITT analysis set comprised randomized subjects.
Measure: Mean (Standard Deviation); unit: points on a score
Arm/Group | Mesalamine | Placebo
Number analyzed (Participants) | 114 | 114
points on a score
  Week 2 | 24.79 (25.92) | 18.75 (33.87)
  Week 4 | 33.58 (29.69) | 28.13 (33.08)
  Week 8 | 34.41 (37.23) | 24.73 (36.42)
Statistical Analysis 1: Comparison: Mesalamine vs Placebo; Change from baseline scores were compared between treatment groups over 8 weeks, at a two-sided 0.05 significance level; Test type: Superiority; p < 0.05, Repeated-measures ANCOVA; Treatment difference = 12.80, 95% CI 2-sided [5.10 to 20.50] — A repeated-measures ANCOVA model with an unstructured correlation matrix was used to calculate estimates

11. Secondary Outcome: Number of Participants Experiencing Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a subject taking part in a clinical trial.
  A 'treatment-emergent AE (TEAE)' is defined as an AE which occurs in the time interval from initial dosing (investigational medicinal product [IMP] intake) to the end of treatment visit.
  Proportion of subjects with any TEAE (serious or non-serious) are presented.
Time Frame: Up to Week 16
Population: The safety analysis set comprised all subjects who received at least 1 dose of IMP, and was analyzed according to actual treatment received.
Measure: Count of Participants; unit: Participants
Groups:
- Mesalamine (Open-Label): Mesalamine 4 g extended release granules (sachet), administered orally QD
Arm/Group | Mesalamine | Placebo | Mesalamine (Open-Label)
Number analyzed (Participants) | 114 | 114 | 170
Participants
  Any TEAE | 28 | 37 | 31
  Serious AE | 1 | 0 | 2

12. Secondary Outcome: Severity of Adverse Events
Description: The proportion of subjects with intensity of AEs (classified as mild, moderate or severe) are presented.
Time Frame: Up to Week 16
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamine | Placebo | Mesalamine (Open-Label)
Number analyzed (Participants) | 114 | 114 | 170
Participants
  Mild | 23 | 27 | 21
  Moderate | 6 | 15 | 11
  Severe | 5 | 3 | 1

13. Secondary Outcome: Proportion of Subject With Abnormal Laboratory Values (Hematology)
Description: Proportion of subjects with markedly abnormal changes from baseline in hematology values are presented.
  >= greater than equal to; <= less than equal to.
Time Frame: Up to Week 16
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamine | Placebo | Mesalamine (Open-Label)
Number analyzed (Participants) | 114 | 114 | 170
Participants
  Eosinophils/Leukocytes (%), Normal>=10 to Abnormal: number analyzed (Participants) | 108 | 108 | 165
  Eosinophils/Leukocytes (%), Normal>=10 to Abnormal | 0 | 2 | 4
  Erythrocytes (10^6/uL), Low<=3.5 to Abnormal: number analyzed (Participants) | 10 | 11 | 15
  Erythrocytes (10^6/uL), Low<=3.5 to Abnormal | 2 | 4 | 4
  Erythrocytes (10^6/uL), Normal<=3.5 to Abnormal: number analyzed (Participants) | 101 | 98 | 153
  Erythrocytes (10^6/uL), Normal<=3.5 to Abnormal | 1 | 0 | 2
  Hematocrit (%), Low<=0.32 to Abnormal: number analyzed (Participants) | 13 | 11 | 20
  Hematocrit (%), Low<=0.32 to Abnormal | 4 | 1 | 5
  Hematocrit (%), Normal<=0.32 to Abnormal: number analyzed (Participants) | 98 | 98 | 147
  Hematocrit (%), Normal<=0.32 to Abnormal | 0 | 3 | 4
  Hematocrit (%), Normal>=0.56 to Abnormal: number analyzed (Participants) | 98 | 98 | 147
  Hematocrit (%), Normal>=0.56 to Abnormal | 0 | 1 | 0
  Hemoglobin (g/dL), Low<=115 to Abnormal: number analyzed (Participants) | 35 | 35 | 53
  Hemoglobin (g/dL), Low<=115 to Abnormal | 21 | 23 | 37
  Hemoglobin (g/dL), Normal<=115 to Abnormal: number analyzed (Participants) | 78 | 75 | 117
  Hemoglobin (g/dL), Normal<=115 to Abnormal | 12 | 15 | 29
  Leukocytes (10^3/uL), Normal <=2.8 to Abnormal: number analyzed (Participants) | 103 | 104 | 155
  Leukocytes (10^3/uL), Normal <=2.8 to Abnormal | 1 | 0 | 2
  Leukocytes (10^3/uL), Normal >=16.0 to Abnormal: number analyzed (Participants) | 103 | 104 | 155
  Leukocytes (10^3/uL), Normal >=16.0 to Abnormal | 0 | 2 | 2
  Leukocytes (10^3/uL), High >=16.0 to Abnormal: number analyzed (Participants) | 8 | 5 | 12
  Leukocytes (10^3/uL), High >=16.0 to Abnormal | 0 | 1 | 1
  Lymphocytes/Leukocytes (%), Low<=10 to Abnormal: number analyzed (Participants) | 22 | 25 | 35
  Lymphocytes/Leukocytes (%), Low<=10 to Abnormal | 0 | 3 | 1
  Lymphocytes/Leukocytes (%), Normal<=10 to Abnormal: number analyzed (Participants) | 90 | 84 | 133
  Lymphocytes/Leukocytes (%), Normal<=10 to Abnormal | 4 | 2 | 6
  Lymphocytes/Leukocytes (%), High>=80 to Abnormal: number analyzed (Participants) | 1 | 1 | 2
  Lymphocytes/Leukocytes (%), High>=80 to Abnormal | 1 | 0 | 1
  Neutrophils/Leukocyte (%), Normal<=15 to Abnormal: number analyzed (Participants) | 98 | 93 | 148
  Neutrophils/Leukocyte (%), Normal<=15 to Abnormal | 2 | 0 | 2
  Neutrophils/Leukocyte (%), Normal>=90 to Abnormal: number analyzed (Participants) | 98 | 93 | 148
  Neutrophils/Leukocyte (%), Normal>=90 to Abnormal | 0 | 1 | 2
  Neutrophils/Leukocyte (%), High >=90 to Abnormal: number analyzed (Participants) | 15 | 17 | 22
  Neutrophils/Leukocyte (%), High >=90 to Abnormal | 0 | 1 | 1
  Platelets (10^3/uL), High>=700 to Abnormal: number analyzed (Participants) | 19 | 22 | 34
  Platelets (10^3/uL), High>=700 to Abnormal | 2 | 0 | 2

14. Secondary Outcome: Proportion of Subjects With Abnormal Laboratory Values (Coagulation)
Description: Proportion of subjects with markedly abnormal changes from baseline values in coagulation laboratory values are presented.
  INR= International normalized ratio.
Time Frame: Up to Week 16
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamine | Placebo | Mesalamine (Open-Label)
Number analyzed (Participants) | 114 | 114 | 170
Participants
  Prothrombin INR, Normal <0.8 to Abnormal: number analyzed (Participants) | 81 | 80 | 127
  Prothrombin INR, Normal <0.8 to Abnormal | 0 | 0 | 1
  Prothrombin INR, Normal >1.1 to Abnormal: number analyzed (Participants) | 81 | 80 | 127
  Prothrombin INR, Normal >1.1 to Abnormal | 14 | 14 | 28
  Prothrombin INR, High >1.1 to Abnormal: number analyzed (Participants) | 20 | 22 | 40
  Prothrombin INR, High >1.1 to Abnormal | 4 | 10 | 22

15. Secondary Outcome: Proportion of Subjects With Abnormal Laboratory Values (Serum Chemistry)
Description: Proportion of subjects with markedly abnormal changes in serum chemistry laboratory values are presented.
  ALT= Alanine aminotransferase; AST= Aspartate aminotransferase; BUN= Blood urea nitrogen; GGT= Gamma glutamyl transferase.
Time Frame: Up to Week 16
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamine | Placebo | Mesalamine (Open-Label)
Number analyzed (Participants) | 114 | 114 | 170
Participants
  ALT (U/L), Normal >3xULN to Abnormal: number analyzed (Participants) | 110 | 108 | 169
  ALT (U/L), Normal >3xULN to Abnormal | 1 | 0 | 2
  AST (U/L), Normal >3xULN to Abnormal: number analyzed (Participants) | 107 | 107 | 163
  AST (U/L), Normal >3xULN to Abnormal | 1 | 0 | 2
  AST (U/L), High >3xULN to Abnormal: number analyzed (Participants) | 5 | 5 | 7
  AST (U/L), High >3xULN to Abnormal | 0 | 0 | 1
  Bilirubin (mg/dL), Normal >=1.5xULN to Abnormal: number analyzed (Participants) | 106 | 100 | 157
  Bilirubin (mg/dL), Normal >=1.5xULN to Abnormal | 1 | 0 | 1
  Bilirubin (mg/dL), High >=1.5xULN to Abnormal: number analyzed (Participants) | 7 | 10 | 13
  Bilirubin (mg/dL), High >=1.5xULN to Abnormal | 2 | 1 | 4
  BUN (mg/dL), Normal >=10.7 to Abnormal: number analyzed (Participants) | 102 | 92 | 145
  BUN (mg/dL), Normal >=10.7 to Abnormal | 0 | 1 | 1
  Calcium (mg/dL), Normal <=1.8 to Abnormal: number analyzed (Participants) | 110 | 104 | 162
  Calcium (mg/dL), Normal <=1.8 to Abnormal | 1 | 0 | 1
  Chloride (mmol/L), Normal >=115 to Abnormal: number analyzed (Participants) | 94 | 98 | 146
  Chloride (mmol/L), Normal >=115 to Abnormal | 1 | 0 | 1
  Chloride (mmol/L), High >=115 to Abnormal: number analyzed (Participants) | 18 | 12 | 23
  Chloride (mmol/L), High >=115 to Abnormal | 1 | 0 | 1
  GGT (U/L), High >3xULN to Abnormal: number analyzed (Participants) | 13 | 10 | 16
  GGT (U/L), High >3xULN to Abnormal | 2 | 2 | 4
  Glucose (mg/dL), Normal >=10 to Abnormal: number analyzed (Participants) | 94 | 85 | 134
  Glucose (mg/dL), Normal >=10 to Abnormal | 1 | 1 | 1
  Glucose (mg/dL), High >=10 to Abnormal: number analyzed (Participants) | 13 | 20 | 25
  Glucose (mg/dL), High >=10 to Abnormal | 0 | 2 | 1
  Potassium (mmol/L), Normal <=3.0 to Abnormal: number analyzed (Participants) | 107 | 110 | 166
  Potassium (mmol/L), Normal <=3.0 to Abnormal | 1 | 0 | 1
  Potassium (mmol/L), Normal >=5.8 to Abnormal: number analyzed (Participants) | 107 | 110 | 166
  Potassium (mmol/L), Normal >=5.8 to Abnormal | 1 | 0 | 3
  Potassium (mmol/L), High >=5.8 to Abnormal: number analyzed (Participants) | 5 | 2 | 3
  Potassium (mmol/L), High >=5.8 to Abnormal | 0 | 0 | 1
  Sodium (mmol/L), Low<=130 to Abnormal: number analyzed (Participants) | 1 | 1 | 1
  Sodium (mmol/L), Low<=130 to Abnormal | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: TEAE occurred in the time interval from initial dosing (IMP intake) to the end of trial visit, up to 8 weeks for the Mesalamine and Placebo Arms and an additional 8 weeks for the Open-Label extension period.
Description: TEAEs were defined as AE which occurred in the time interval from initial dosing (IMP intake) to the end of treatment visit.
Arm/Group | Mesalamine | Placebo | Mesalamine (Open-Label)
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/114 | 0/170
Serious Adverse Events (participants affected / at risk) | 1/114 | 0/114 | 2/170
Other Adverse Events (participants affected / at risk) | 19/114 | 13/114 | 8/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesalamine (N=114) | Placebo (N=114) | Mesalamine (Open-Label) (N=170)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesalamine (N=114) | Placebo (N=114) | Mesalamine (Open-Label) (N=170)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 3 (3) | 10 (10) | 4 (4)
C-reactive protein increased (Investigations) | 6 (6) | 1 (1) | 0 (0)
Faecal calprotectin increased (Investigations) | 5 (5) | 2 (2) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (2):
  • Study Protocol (2017-01-11): https://cdn.clinicaltrials.gov/large-docs/67/NCT02522767/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT02522767/SAP_001.pdf